CLINICAL TRIAL: NCT06596031
Title: Health Coaching in Addition to a Digital Resource to Promote Self-management for Patients Waiting for Total Hip or Knee Replacements: A Randomised Feasibility Trial
Brief Title: Health Coaching for Patients Waiting for Total Hip or Knee Replacements
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ER68359613
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Arthritis Knee; Arthritis of Hip
Keywords: joint replacement surgery; digital resource; health coaching; telehealth; self management

STUDY DESIGN:
Intervention Model Description: Pilot study of a single-blinded, randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health coaching (Experimental): Participants randomized to the intervention group will receive access to the Active Wait program, which includes remote, self-paced (asynchronous) education, exercise, and nutritional advice delivered via a web-based platform. The participants in the intervention group will have access to the program, in conjunction with health coaching.
  Patients undertaking health coaching will be assigned a personal health coach who will provide support to increase their ability to self-manage through self- regulation principles of behaviour change. Health coaching sessions will be delivered remotely (via telephone or video conferencing) a maximum of 8-times during a 12-week intervention period. Sessions are limited to 1 hour, offering education, self-management strategies, barrier and facilitator identification, support and encouragement, goal setting, action planning and self-monitoring with the intention to facilitate positive and sustainable lifestyle and behaviour changes.
  Interventions: Behavioral: Health coaching
- Digital toolkit (Active Comparator): Patients in the active-comparator group will be given a link to the same Digital Toolkit. The digital toolkit is a 12-week non-contact programme titled Active Wait, which offers education, self-management techniques and an unsupervised strength programme. The website Active Wait can be accessed via the link: https://protect-au.mimecast.com/s/8_5gCP7yRZiWn3q3FzwqnS?domain=sheffieldachesandpains.com/
  Interventions: Behavioral: Digital toolkit

INTERVENTIONS:
Behavioral: Health coaching — The core belief in coaching is that people are resourceful and that the participant knows what is best for themselves. If the participants are assigned to the health coaching group, they will have access to a health coach with a physiotherapist background. Instead of offering physiotherapy advice, however, the health coaching will work with the participant to come up with ideas that work the best for them to manage their health and wellness to prepare for surgery, including addressing some difficulties the participant are facing when using the online resource.
  Arms: Health coaching
Behavioral: Digital toolkit — This intervention provides, via a website, self-management support of preoperative rehabilitation for hip or knee replacement based on NICE guidelines Joint replacement (primary): hip and knee. This includes guidance for patients to undertake a strengthening programme that will aid recovery, lifestyle behaviours including weight management, diet and smoking cessation, and maximising functional independence and quality of life before surgery.
  Arms: Digital toolkit

SUMMARY:
This pilot study aims to evaluate the feasibility of collecting objective data on physical performance to measure the impact of health coaching in addition to a digital resource (Active Wait) and enable sample size calculation for a larger scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled on the waitlist for a total joint replacement surgery for hip/knee, ie clinically and radiographically diagnosed, symptomatic knee/hip osteoarthritis deemed suitable for surgical intervention;
* have access to the internet and the ability to navigate web-based programs;
* able and willing to travel to Advanced Wellbeing Research Centre for baseline and follow-up assessments;
* able to comprehend the requirements and purpose of the study and give informed consent

Exclusion Criteria:

* other musculoskeletal lower limb or back conditions requiring assessment or treatment by a health professional in the last 6 months;
* neurological impairment or condition affecting lower limb function; conditions listed as both absolute and relative contraindications for physical activities by the American College of Sports Medicine (ACSM), such as unstable angina, uncontrolled diabetes;
* systemic inflammatory disease (e.g. rheumatoid arthritis);
* previous total joint replacement surgery (hip or knee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Global rating of change | 12 weeks
  Bowens Framework - acceptability (Perceived benefits) 7-point likert scale global rating of change (GROC) with -3 being worse, 0 being no change and 3 being better
Perceived Satisfaction | 12 weeks
  Bowens Framework - acceptability (Perceived satisfaction). How satisfied were you with the overall information, level of support, and ease of use of the program? Measured on a numeric rating scale, where 0 means not satisfied, 10 means significant satisfaction.
Rate of retention | 12 weeks
  Bowens Framework - acceptability, percentage of participants progressing from baseline, to midpoint and post-intervention assessments
Drop out rate | 12 weeks
  Bowens Framework - acceptability, percentage of people discontinuing in both groups
Adverse events | 12 weeks
  Bowens Framework- practicality, measured by number, type and severity of adverse events
Rate of service utilisation | 12 weeks
  Bowens Framework - implementation, measured by the number of attended sessions (health coaching) number of days during the week using the active wait website
Rates of recruitment | 12 weeks
  Bowens Framework - demand, measured by n number of recruitment per week.

SECONDARY OUTCOMES:
Demographics | 12 weeks
  height and weight aggregated to arrive at one reported value BMI, in units kg/m^2
Arthritis Self-Efficacy Scale (ASES-8) | 12 weeks
  Self efficacy questionnaire. Contains 8 items, each measured on a scale from 1-10. Higher score indicates greater self-efficacy.
International physical activity questionnaire-short form (IPAQ-SF) | 12 weeks
  Physical activity level is measured in three categories, walking, moderate-intensity activities, vigorous-intensity activities, in addition to sitting. Their score is then expressed as MET-min per week.
EuroQoL Group's 5-dimension (EQ-5D-5L) | 12 week
  Health related quality of life questionnaire. Each dimension of the EQ-5D has 5 levels from 1-5. 1 indicates full health state, 5 indicates worse the problem. The last question, EQ-5D health scale is a scale between 0-100, where 0 indicates worst health, 100 indicates best health.
Visual Analogue Scale | 12 week
  VAS 10 point scale for self report of pain level. With 1 being no pain and 10 being maximal pain.
Oxford knee/hip score | 12 week
  Joint specific function questionnaire. The questionnaire contains 6 questions. Each question ranges from 0 to 4, with 4 being the best outcome. The highest score is 48.
Knee flexion/extension strength | 12 week
  Biodex for isometric strength testing, peak torque will be calculated in N.m
4 x 10m walk test | 12 week
  The average time taken to complete a 10m lap (s)
12 steps test | 12 week
  Time taken to complete 1 flight of 12 steps (s)
Time up and go | 12 week
  Amount of time taken to complete a lap from sitting to standing, walking for 3 m, turn around a marker and return to sitting position (s)
Sit to stand test | 12 week
  Number of full repetitions from sitting to standing in a 30s period
Minutes in sedentary activities | 1 week baseline and 1 week at completion
  Wearable tracking using ActivPAL

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Wellbeing Research Centre, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a pilot study assessing the feasibility of conducting a larger scale randomised control trial. Limited efficacy is the secondary outcome only.

REFERENCES:
- [Background] Abbott JH, Schmitt J. Minimum important differences for the patient-specific functional scale, 4 region-specific outcome measures, and the numeric pain rating scale. J Orthop Sports Phys Ther. 2014 Aug;44(8):560-4. doi: 10.2519/jospt.2014.5248. Epub 2014 May 14. PMID 24828475
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Lienhard K, Lauermann SP, Schneider D, Item-Glatthorn JF, Casartelli NC, Maffiuletti NA. Validity and reliability of isometric, isokinetic and isoinertial modalities for the assessment of quadriceps muscle strength in patients with total knee arthroplasty. J Electromyogr Kinesiol. 2013 Dec;23(6):1283-8. doi: 10.1016/j.jelekin.2013.09.004. Epub 2013 Sep 23. PMID 24113423
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Lyden K, Keadle SK, Staudenmayer J, Freedson PS. The activPALTM Accurately Classifies Activity Intensity Categories in Healthy Adults. Med Sci Sports Exerc. 2017 May;49(5):1022-1028. doi: 10.1249/MSS.0000000000001177. PMID 28410327
- [Background] Norman R, Cronin P, Viney R. A pilot discrete choice experiment to explore preferences for EQ-5D-5L health states. Appl Health Econ Health Policy. 2013 Jun;11(3):287-98. doi: 10.1007/s40258-013-0035-z. PMID 23649892
- [Background] Sarabon N, Ceh T, Kozinc Z, Smajla D. Adapted protocol of rate of force development and relaxation scaling factor for neuromuscular assessment in patients with knee osteoarthritis. Knee. 2020 Dec;27(6):1697-1707. doi: 10.1016/j.knee.2020.09.023. Epub 2020 Nov 13. PMID 33197807
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Wallis JA, Webster KE, Levinger P, Taylor NF. What proportion of people with hip and knee osteoarthritis meet physical activity guidelines? A systematic review and meta-analysis. Osteoarthritis Cartilage. 2013 Nov;21(11):1648-59. doi: 10.1016/j.joca.2013.08.003. Epub 2013 Aug 12. PMID 23948979
- [Background] Wilcox S, Schoffman DE, Dowda M, Sharpe PA. Psychometric properties of the 8-item english arthritis self-efficacy scale in a diverse sample. Arthritis. 2014;2014:385256. doi: 10.1155/2014/385256. Epub 2014 Aug 21. PMID 25215233